CLINICAL TRIAL: NCT00719524
Title: An Open-label, Non-randomized, Dose Evaluation, Safety and Pharmacokinetics Phase I Study of AVE8062 in Combination With Platinum Salts (Cisplatin or Carboplatin) and Taxanes (Docetaxel or Paclitaxel), Every 3 Weeks, in Patients With Advanced Solid Tumors.
Brief Title: AVE8062 in Combination With Platinum-taxane Doublet in Advanced Solid Tumor
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Sanofi (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TCD10620; EudraCT: 2007-006676-11
Record Dates: First submitted 2008-07-17; First posted 2008-07-21 (Estimated); Last update posted 2013-03-11 (Estimated); Status verified 2013-03

CONDITIONS: Neoplasms
Keywords: Neoplasms; Antineoplastic Combined Chemotherapy Protocol
MeSH Terms: conditions — Neoplasms | interventions — AC 7700

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Experimental)
  Interventions: Drug: OMBRABULIN (AVE8062)

INTERVENTIONS:
Drug: OMBRABULIN (AVE8062) — Dose escalation study with combination chemotherapy

SUMMARY:
The purpose of this study is to determine the recommended dose of the combination of AVE8062 with platinum salts (cisplatin or carboplatin) and taxanes (docetaxel or paclitaxel) in patients with advanced solid tumors for which platinum-taxane doublet constitutes mainstay of care.

ELIGIBILITY:
Inclusion Criteria:

* Advanced neoplastic disease (i.e. metastatic or locally advanced disease) for which platinum-taxane doublet regimens are approved or constitutes the mainstay of care such as non small cell lung cancer, epithelial ovary cancer, gastric cancer, transitional cell and bladder cancer and head and neck cancer.
* Eastern cooperative oncology group (ECOG) performance status of 0 to 1.

Exclusion Criteria:

* Concurrent treatment with any other anticancer therapy, including chemotherapy, immunotherapy, radiotherapy (excluding radiotherapy with palliative intent on non-target lesions), targeted therapy, gene therapy, or patients planning to receive these treatments during the study.
* Absence of histologically or cytologically proven cancer at the first diagnosis.
* Negative serum/urinary pregnancy test
* Washout period of 3 weeks for prior anti-tumor therapy or any investigational treatment

The above information is not intended to contain all considerations relevant to a patient's potential participation in a clinical trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 71 (Actual)
Dates: Start 2008-07; Primary Completion 2013-02 (Actual); Study Completion 2013-02 (Actual)

PRIMARY OUTCOMES:
Recommended dose of the combination based on Dose Limiting Toxicities observed | Cycle 1

SECONDARY OUTCOMES:
Overall safety profile | Treatment period
Pharmacokinetic profile | Cycle 1
Anti-tumor activity of the combination | Every 2 cycles

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Sciences & Operations, Study Director — Sanofi
Locations (3):
- Investigational Site Number 250001, Villejuif, France
- Investigational Site Number 380001, Milan, Italy
- Investigational Site Number 756001, Bellinzona, Switzerland

REFERENCES:
- [Derived] Bahleda R, Sessa C, Del Conte G, Gianni L, Capri G, Varga A, Oprea C, Daglish B, Hospitel M, Soria JC. Phase I clinical and pharmacokinetic study of ombrabulin (AVE8062) combined with cisplatin/docetaxel or carboplatin/paclitaxel in patients with advanced solid tumors. Invest New Drugs. 2014 Dec;32(6):1188-96. doi: 10.1007/s10637-014-0119-0. Epub 2014 Jun 6. PMID 24898305